CLINICAL TRIAL: NCT05096676
Title: Understanding Oxytocin's Neural and Behavioral Effects in Adolescents Diagnosed With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Ilanit gordon (Other)
Responsible Party: Sponsor-Investigator, Prof. Ilanit gordon, Principal Investigator, Bar-Ilan University, Israel
Organization: Bar-Ilan University, Israel (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16082021IG
Record Dates: First submitted 2021-08-16; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Autism Spectrum Disorder; Oxytocin
Keywords: Autism; MEG; Social perception
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Youth with autism participated in a randomized, double-blind placebo-controlled trial. Participants visited the lab for two sessions. In one of the sessions, they received oxytocin, and in the other, they received the placebo. Intranasal doses of 40 international units of oxytocin (IU)/mL were prepared by the "Maayan-Haim" pharmacy, Israel. We used age-dependent dosing such that participants aged 13-18 years received a dose of 24 IU (3 puffs to each nostril), and younger participants (aged 12 years) received 16 IU. Typically-developing youth underwent the same experimental procedure but did not receive oxytocin or placebo due to ethical constraints in Israel.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adolescents diagnosed with Autism spectrum disorder (Experimental): Participants in the ASD group received oxytocin and placebo in a randomized, double-blind placebo-controlled manner.
  Interventions: Drug: Oxytocin: Including placebo
- Typically developing adolescents (No Intervention): Control participants were recruited using online ads. This group did not receive oxytocin or placebo due to ethical constraints in Israel.

INTERVENTIONS:
Drug: Oxytocin: Including placebo — Individual received age-dependent dosing of oxytocin and placebo. Participants aged 13-18 years received a dose of 24 IU (3 puffs to each nostril), and younger participants (aged 12 years) received 16 IU.
  Arms: Adolescents diagnosed with Autism spectrum disorder

SUMMARY:
The investigators explored the neural and behavioral effect of oxytocin on youth with Autism spectrum disorder using magnetoencephalography (MEG). The investigators hypothesize that oxytocin will modulate neural activity to resemble patterns observed in the age-matched control group.

Thirty-two adolescents with autism and 26 typically developing adolescents participated in this randomized, double-blind MEG study. Individuals with autism arrived at the lab twice and received an acute dose of intranasal oxytocin or placebo in each session. During the scans, participants were asked to complete several tasks related to social perception - such as identification of social and non-social stimuli.

DETAILED DESCRIPTION:
In the current study, the investigators aimed to explore oxytocin's influences on neural components that relate to social processing. Namely, we focused on M100, M170, and M250, which tend to show atypical patterns in individuals with autism.

The investigators also examined the effects of oxytocin on time dynamics - the change in specific oscillation over time and its effects on neural connectivity patterns.

ELIGIBILITY:
Inclusion Criteria:

* Males, aged 12-18 years
* Native Hebrew speakers
* Normal or corrected-to-normal vision
* Participants in the ASD group had to meet the criteria for ASD in the diagnostic and statistical manual of mental disorders (DSM-5)

Exclusion Criteria:

* Chronic medical problems
* Cardiovascular risk factors
* CNS disease
* Other mental illnesses
* Use of prohibited medications
* Mental retardation
* Impaired vision
* Impaired hearing
* History of significant head injury or neurological illness
* Current substance dependence diagnosis
* Metallic implants, braces or devices in the body

Ages: 12 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
The change in social-related neural components (time-locked neural activity) with and without oxytocin | During each session
  The amplitude (tesla) of three social related neural components will be measured using MEG device

SECONDARY OUTCOMES:
The change in oscillatory activity - power magnitude of Delta, Theta, Alpha, Beta and Gamma neural bands with and without oxytocin | During each session
  The overall power of neural oscillatory activity will be measured using MEG device
The change in behavioral measurments - reaction times and accurecy rates, with and without oxytocin | During each session
  Reaction times will be measured in milliseconds and accurecy rates will be defined as the percentage of correct responses

REFERENCES:
- [Derived] Korisky A, Goldstein A, Gordon I. The dual neural effects of oxytocin in autistic youth: results from a randomized trial. Sci Rep. 2022 Sep 29;12(1):16304. doi: 10.1038/s41598-022-19524-7. PMID 36175473
- [Derived] Korisky A, Gordon I, Goldstein A. Oxytocin impacts top-down and bottom-up social perception in adolescents with ASD: a MEG study of neural connectivity. Mol Autism. 2022 Sep 5;13(1):36. doi: 10.1186/s13229-022-00513-6. PMID 36064612

DOCUMENTS (1):
  • Statistical Analysis Plan (2015-10-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT05096676/SAP_000.pdf